CLINICAL TRIAL: NCT05609565
Title: Hybrid Anesthesia for Ambulatory Knee Arthroscopy Using Intrathecal Prilocaine and Adductor Canal Block vs Intrathecal Bupivacaine Alone: a Randomized Controlled Trial
Brief Title: Intrathecal Prilocaine and Adductor Canal Block vs Intrathecal Bupivacaine Alone for Ambulatory Knee Arthroscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ibrahim Mamdouh Esmat, Assistant Professor of Anesthesia and Intensive Care Department, Faculty of Medicine, Ain- shams University, Cairo, Egypt., Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FMASU MS 706/ 2022
Record Dates: First submitted 2022-11-03; First posted 2022-11-08 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Anesthesia, Spinal; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator)
  Interventions: Drug: spinal anesthesia with hyperbaric prilocaine+adductor canal block (ACB) with bupivacaine
- Group 2 (Active Comparator)
  Interventions: Drug: spinal anesthesia with bupivacaine

INTERVENTIONS:
Drug: spinal anesthesia with hyperbaric prilocaine+adductor canal block (ACB) with bupivacaine — spinal anesthesia with hyperbaric prilocaine+adductor canal block (ACB) with bupivacaine
  Arms: Group 1
Drug: spinal anesthesia with bupivacaine — spinal anesthesia with bupivacaine
  Arms: Group 2

SUMMARY:
- Although bupivacaine is safe and has a low rate of transient neurologic symptoms, the prolonged sensory and motor block is a drawback for day-case spinal anesthesia.Intrathecal hyperbaric prilocaine causes a much shorter motor block, with a similar onset time and lower inter-individual variability in motor block duration. Furthermore, the peripheral nerve block is used as an adjunct to the spinal anesthesia to prolong the surgical anesthetic conditions.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) score I-II.
* Body mass index < 35 kg/m2

Exclusion Criteria:

* Patient's refusal.
* Known coagulopathy.
* Known peripheral neuropathy or neurological deficits.
* Known allergy to study drugs.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
The duration of motor block (minutes) | 24 hours postoperatively
  The duration of motor block (minutes)

CONTACTS AND LOCATIONS:
Locations (1):
- Ain-Shams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No